CLINICAL TRIAL: NCT01563016
Title: Glucose as a Mediator of Self-control Performances in Patients With Schizophrenia: A Randomized Controlled Study
Brief Title: Glucose as a Mediator of Self-control Performances in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: selfcontrolvsglucose
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Schizophrenia
Keywords: schizophrenia; Psychotic Disorders; Psychoses
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Glucose & Depleting (Experimental): participants will perform in a depleting task and receive a glucose drink
  Interventions: Dietary Supplement: glucose drink
- Glucose & non-depleting (Placebo Comparator): participants will perform in a non-depleting task and receive a glucose drink
  Interventions: Dietary Supplement: glucose drink
- Placebo & depleting (No Intervention): participants will perform in a depleting task and receive a placebo drink
- Placebo & non depleting (No Intervention): participants will perform in a non depleting task and receive a placebo drink

INTERVENTIONS:
Dietary Supplement: glucose drink — participants will receive a drink rich in glucose
  Arms: Glucose & Depleting; Glucose & non-depleting

SUMMARY:
The research aims to investigate the relationship between self-control ability and blood glucose level in schizophrenic patients. The main purpose of the present study is to explore whether the close relationship of blood glucose and self-regulatory strength observed in healthy individuals, is applicable to schizophrenic patients. More specifically, the current study aims

* to investigate whether the exertion of self-control reduces blood glucose,
* to examine whether low level of blood glucose deteriorates subsequent self-control performances
* to examine whether restoring the glucose level eliminates these impairments, in schizophrenic patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 or above
* DSM-IV diagnosis of schizophrenia, schizoaffective disorder, schizophreniform psychosis, brief psychosis, psychosis NOS or delusional disorder
* Cantonese-speaking Chinese
* Ability to understand the nature of the study and sign informed consent

Exclusion Criteria:

* Organic Brain disorder
* Known history of intellectual disability
* Priority Follow Up (Subtarget or Target)
* All allergic to any sugar or artificial sweeteners
* Diabetics
* Physical Disability

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Blood Glucose Level | baseline, after depleting task
self control tasks (handgrip, stroop, figure tracing task) | after 12-minutes metabolizing phase

CONTACTS AND LOCATIONS:
Overall Officials: Eric YH Chen, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, China